CLINICAL TRIAL: NCT06683846
Title: Ivonescimab (PD-1/VEGF Bispecpecial Antibody) in the Treatment of Multiple Advanced Tumors: a Multi-cohort, Multi-center, Single-arm Phase II Study
Brief Title: Ivonescimab in the Treatment of Multiple Advanced Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Hongxia Wang, Director of oncology department, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK112-US-01
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Pheochromocytoma/Paraganglioma; Rhabdomyosarcoma; Paget Disease, Extramammary; Renal Angiomyolipoma; Perivascular Epithelioid Cell Tumor, Malignant; Sarcoma; Urachal Cancer; Neuroendocrine Cancer; Basal Cell Carcinomas; Sarcomatoid Carcinoma; Penile Cancer; Adrenal Cortical Cancer; Germ Cell Cancer Metastatic; Non-Clear Cell Renal Cell Carcinoma; Prostate Cancers; Clear Cell Renal Cancer; Urothelial Carcinoma; Kidney Cancer; Rare Tumors
Keywords: rare tumor; Ivocizumab; immunotherapy
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma; Rhabdomyosarcoma; Paget Disease, Extramammary; Angiomyolipoma; Perivascular Epithelioid Cell Neoplasms; Sarcoma; Urachal cancer; Carcinoma, Neuroendocrine; Carcinoma, Basal Cell; Carcinoma; Penile Neoplasms; Prostatic Neoplasms; Carcinoma, Transitional Cell; Kidney Neoplasms

STUDY DESIGN:
Intervention Model Description: single-arm, multi-cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ivonescimab (20mg/kg）in rare tumors (Experimental): Participants will receive Ivonescimab 20mg/kg of body weight via intravenous (IV) infusion on Days 1 of a 21-day treatment cycle until disease progression or unacceptable toxicity, or full 2 years of treatment, whichever occurs first.
  Interventions: Drug: Ivocizumab

INTERVENTIONS:
Drug: Ivocizumab — Administered via intravenous (IV) infusion

SUMMARY:
The goal of this clinical trial is to learn if Ivonescimab works to treat advanced rare tumors including cohort 1: PAGET's disease of scrotum with infiltrating sweat gland carcinoma. cohort 2: Metastatic paraganglioma and pheochromocytoma. cohort 3: Metastatic renal angiomyolipoma and malignant perivascular epithelioid cell tumor.

cohort 4: Rhabdomyosarcoma and Ewing's sarcoma cohort 5: Collecting duct carcinoma cohort 6: Urachal carcinoma. cohort 7: Neuroendocrine cancer. cohort 8: Basal cell carcinoma and sarcomatoid carcinoma. cohort 9: Penile cancer. cohort 10: Adrenal cortical cancer. cohort 11: Metastatic germ cell tumors, failure of standard cisplatin based therapy (mostly testicular cancer).

cohort 12: Non-clear cell renal carcinoma (including renal papillary renal carcinoma); Renal cancer cannot be classified).

cohort 13: Non-clear cell renal carcinoma (including chromophobe renal carcinoma) cohort 14: Other rare tumors that cannot be classified (such as testicular reticulum adenocarcinoma, etc.).

cohort 15: Prostate cancer. cohort 16: Clear cell renal carcinoma. (16.1: received PD-1; 16.2: no PD-1 received) cohort 17: Urothelial carcinoma. cohort 18: Kidney cancer with brain metastases. cohort 19: Brain metastases of urothelial carcinoma. cohort 20: Rare tumors with brain metastases.

It will also learn about the safety of Ivonescimab. The main questions it aims to answer are:

Does Ivonescimab improve the objective response rate and prolong the survival of participants? What medical problems do participants have when taking Ivonescimab?

Participants will:

Receive Ivonescimab 20mg/kg intravenously every 21 days until disease progression, intolerable toxicity, or full 2 years of treatment, whichever occurs first.

Be performed imaging evaluation according to RECIST 1.1 every 9 weeks for 1 year of treatment and every 12 weeks after 1 year Be recorded any adverse events in the whole study period including type, incidence, grade, severity, duration, and association with the study drug according to NCI-CTCAE V5.0 criteria

DETAILED DESCRIPTION:
This is a prospective, multi-cohort phase II study. Primary objectives is to evaluate the objective response rate (ORR) of Ivonescimab in the treatment of multiple rare advanced tumors. Secondary objectives is to evaluate the imaging progression-free survival (PFS), overall survival (OS), quality of life (QoL), and safety in the treatment of multiple rare advanced tumors with Ivonescimab.

A total of 20 cohorts were included:

cohort 1: PAGET's disease of scrotum with infiltrating sweat gland carcinoma. cohort 2: Metastatic paraganglioma and pheochromocytoma. cohort 3: Metastatic renal angiomyolipoma and malignant perivascular epithelioid cell tumor.

cohort 4: Rhabdomyosarcoma and Ewing's sarcoma cohort 5: Collecting duct carcinoma cohort 6: Urachal carcinoma. cohort 7: Neuroendocrine cancer. cohort 8: Basal cell carcinoma and sarcomatoid carcinoma. cohort 9: Penile cancer. cohort 10: Adrenal cortical cancer. cohort 11: Metastatic germ cell tumors, failure of standard cisplatin based therapy (mostly testicular cancer).

cohort 12: Non-clear cell renal carcinoma (including renal papillary renal carcinoma); Renal cancer cannot be classified).

cohort 13: Non-clear cell renal carcinoma (including chromophobe renal carcinoma) cohort 14: Other rare tumors that cannot be classified (such as testicular reticulum adenocarcinoma, etc.).

cohort 15: Prostate cancer. cohort 16: Clear cell renal carcinoma. (16.1: received PD-1; 16.2: no PD-1 received) cohort 17: Urothelial carcinoma. cohort 18: Kidney cancer with brain metastases. cohort 19: Brain metastases of urothelial carcinoma. cohort 20: Rare tumors with brain metastases. Sample size: using one stage binomial design with power 80% and unilateral alpha value 0.1, it is expected that less than 5% will be ineffective, while 20% will be effective. Considering 10% loss of follow-up, 19 cases will be required. Calculate 20 people per cohort. A total of 400 patients were enrolled.

The study included a screening period (participants signed informed consent no more than 28 days before the first treatment in the study), a treatment period (treatment termination was defined as termination of treatment for any reason, such as imaging confirmation of disease progression, failure to tolerate adverse effects after dose adjustment, or early withdrawal for any reason), and a follow-up period (including end-of-treatment visits, safety visits, and survival follow-up).

Screening period: Participants are required to undergo a screening period within 28 days prior to the study's first treatment to determine eligibility.

Duration of treatment: Patients were treated with ebraxizumab (20mg/kg Q3W every 3 weeks) until disease progression or intolerability of toxicity, or ebraxizumab for 2 years. Reviews were performed every 9 weeks for 1 year of treatment and every 12 weeks after 1 year.

Follow-up period: The safety follow-up period began after the last study treatment, and was followed up once on the 30th day (±7 days). Subjects should go to the research center for the examination of vital signs, physical examination, laboratory examination and other protocol requirements, and evaluate AE, concomitant medication and concomitant treatment.

After the end of the safety follow-up period, the subjects entered the 1-year survival follow-up period, which was conducted every 3 months. They could be visited by telephone follow-up and other effective ways to collect survival information and follow-up treatment information. Survival follow-up lasted until death, loss of follow-up, withdrawal of informed consent, or investigator termination of the study.

Administration regimen: Ivonescimab (AK112), 20mg/kg, 21 days in a cycle, with not less than 90 minutes (±10 minutes) of intravenous infusion, the infusion time can be extended to a maximum of 240 minutes, continuous administration until disease progression, intolerable toxicity, or 2 years of treatment.

Dose adjustment of AK112 is not permitted during treatment, but delayed dosing is permitted for up to 12 weeks (since the last dosing time) if AK112 is discontinued for more than 12 weeks due to glucocorticoid administration for irAE, or if there is an AE that may be unrelated or unrelated to AK112 due to treatment. In both cases that led to the suspension of AK112 for more than 12 weeks, the investigators determined that the patient would benefit from continued treatment and could be allowed to delay treatment for more than 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Individuals able to understand and give written informed consent.
* Histologically or cytologically confirmed cancer of one of the following types:

PAGET's disease of scrotum with infiltrating sweat gland carcinoma Paraganglioma Pheochromocytom, Renal angiomyolipoma Malignant perivascular epithelioid cell tumor, Rhabdomyosarcom Other sarcoma rather than rhabdomyosarcom

* Stage IV disease
* Adequate performance status (ECOG 0-2)
* Expected survival ≥ 3 months.
* Measurable disease by CT or MRI, Or lesions with skin infiltration.
* Adequate hematology without ongoing transfusional support (hemoglobin > 9 g/dL, absolute neutrophil count (ANC) > 1,500 per mm^3, platelets > 100,000 per mm^3).
* Adequate renal and hepatic function (creatinine ≤ 2.0 x institutional upper limit of normal (IULN), bilirubin ≤ 1.5 IULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 x IULN or 5 x IULN if know liver metastases).
* Adequate coagulation function: International Normalized Ratio (INR) ≤1.5 /PT≤1.5×ULN, aPTT≤1.5×ULN.
* Willing to use a medically approved contraceptive method from the enrollment to at least 120 days after the end of the study, and sperm donation to another person or cryopreservation for fertilization and reproduction is not permitted during this period.
* Ability to comply with research visit schedules and other protocol requirements.

Exclusion Criteria:

* With any severe and/or uncontrolled disease. Including: (1)Poor blood pressure control (systolic blood pressure ≥150mmHg or diastolic blood pressure ≥100mmHg); (2) poor control of diabetes (fasting blood sugar [FBG] >10mmol/L);

  ≥2 grade myocardial ischemia or myocardial infarction, arrhythmia (QTc≥470ms), and ≥2 grade congestive heart failure (NYHA classification); (3)active or uncontrolled severe infections requiring systemic antibacterial, antifungal, or antiviral treatment (≥CTCAE 2-level infection), including tuberculosis infection; A history of active tuberculosis; (4)Uncontrolled ascites, pleural effusion, or pericardial effusion that require repeated drainage;
* With active hepatitis (transaminase levels not meeting inclusion criteria; HBV reference: HBV DNA≥2000 IU/ml or ≥10^4 copies/ml; HCV reference: HCV RNA≥2000 IU/ml or ≥10^4 copies/ml; after nucleoside analog antiviral therapy below the above standard, can be included; chronic hepatitis B virus carrier, HBV DNA<10^4 IU/ml, must be treated with antiviral drugs during the trial period to be eligible for enrollment);
* History of immunodeficiency, including HIV positive or subjects with other acquired or congenital immunodeficiency diseases;
* Active autoimmune disease requiring systemic treatment within the past two years, or subjects with an autoimmune disease that the investigator judges may recur or is planned for treatment; except: non-systemic treatment of skin diseases (e.g. vitiligo, alopecia, psoriasis or eczema); autoimmune thyroiditis-induced hypothyroidism requiring stable dose replacement therapy with hormones; 13. Subjects who have experienced severe hypersensitivity reactions after using monoclonal antibodies; individuals who are known to be allergic to the active ingredients or excipients of the study drug;
* Have participated or are currently participating in another clinical study within the past 4 weeks prior to study entry;
* Received a live vaccine within the past 30 days prior to the first dose or plan to receive a live vaccine during the study;
* History of severe allergies;
* At risk of bleeding, or with impaired coagulation function, or currently receiving thrombolytic therapy;
* History of substance abuse with an inability to abstain or a history of mental illness;
* Subjects who, in the opinion of the investigator, have a serious underlying condition that would endanger the subject's safety or impair the subject's ability to complete the study, or who, in the opinion of the investigator, have other reasons not to be enrolled; Subjects who have a history of a clearly defined neurological or psychiatric disorder, such as dementia, epilepsy, or a history of seizure susceptibility;
* Subjects who, in the opinion of the investigator, have a serious underlying condition that would endanger the subject's safety or impair the subject's ability to complete the study (such as severe diabetes, thyroid disorders, and mental illness), or who have a serious and/or unstable medical, psychological, or other condition (including laboratory abnormalities) that would affect the subject's safety or the subject's ability to provide informed consent, or who have any condition that would affect the study protocol and follow-up plan, including psychological, familial, social, or geographic factors;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 12 weeks
  ORR was defined as the proportion of patients who achieved either a complete response (CR) or a partial response (PR) based on the investigator's assessment (RECIST v1.1) that was confirmed by a subsequent scan ≥4 weeks after initial CR/PR.

SECONDARY OUTCOMES:
Progression-free survival(PFS) | 1 year
  PFS was defined as the time between the enrollment and either RECIST1.1-defined progressive disease or death due to any cause, whichever occurred first.
Overall survival (OS) | 2 years
  OS was defined as the time between the enrollment and death due to any cause.
Patient-Reported Quality-of-Life(QoL) | 1 year
  Patient-Reported QoL was evaluated according to the European Organization for Research and Treatment of Cancer QOL Core Questionnaire 30 (EORTC QLQ-30) questionaire.

CONTACTS AND LOCATIONS:
Overall Officials: Hongxia Wang, Doctor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No